CLINICAL TRIAL: NCT01570660
Title: Effects of Glimepiride Monotherapy Versus Combined Neteglinide-Pioglitazone Therapy on Insulin Sensitivity in Type 2 Diabetic Patients
Brief Title: Phielix et al.: Hepatic Fat Content and Adipokines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Diabetes Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 026/2002; 26/2002 (Registry Identifier: Ethikkommisson)
Record Dates: First submitted 2012-03-14; First posted 2012-04-04 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- control group (No Intervention): parallel group without intervention
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — 12 weeks of pioglitazone treatment

SUMMARY:
Thiazoledinediones decrease blood glucose by their insulin-sensitizing properties. Here the investigators examined whether pioglitazone (PIO) improves insulin sensitivity independently of glycemic control and whether adipokines or non-esterfied fatty acids (NEFA) serve as mediators.

ELIGIBILITY:
Inclusion Criteria:

* well controlled patients with type 2 diabetes (Hb1Ac < 8%)
* no insulin therapy
* no co-morbidities
* stable medication use for the last 6 months
* stable body weight the last 6 months
* no diet in the last 6 months

Exclusion Criteria:

* Hb1Ac > 8%
* insulin therapy
* diabetes-related co-morbidities, like cardiovascular disease, neuropathology
* unstable medication use
* unstable body weight in the last 6 months (> 5 kg)
* following a diet in the last 6 months

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2002-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
whole body insulin sensitivity | within a minimal of 1 week before the start of the 12 weeks pioglitazone or glimepiride treatment and after the last day of the treatment period.
  Participants underwent a two-step hyperinsulinemic euglycemic clamp to determine insulin sensitivity, expressed as rate of glucose disposal (Rd) in mg/kg/min.

SECONDARY OUTCOMES:
intrahepatocellular lipid content | within a minimal of 1 week before the start of the 12 weeks pioglitazone or glimepiride treatment and after the last day of the treatment period.
  Liver proton-magnetic resonance spectroscopy was applied to determine liver fat (HCL) in % (relative to the water peak).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Prof., Principal Investigator — Institute for Clinical Diabetology, German Diabetes Center, D-40225, Düsseldorf, Germany; Division of Endocrinology and Metabolism, Department of Internal Medicine III, Medical University of Vienna, Vienna, Austria. Department of Metabolic Diseases, Un
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Phielix E, Brehm A, Bernroider E, Krssak M, Anderwald CH, Krebs M, Schmid AI, Nowotny P, Roden M. Effects of pioglitazone versus glimepiride exposure on hepatocellular fat content in type 2 diabetes. Diabetes Obes Metab. 2013 Oct;15(10):915-22. doi: 10.1111/dom.12112. Epub 2013 May 1. PMID 23574533